CLINICAL TRIAL: NCT03711591
Title: Proximal Humerus Fixation With the Conventus Cage™ PH Device A Post-Approval Observational Data Collection Study, A Single-Center Study, Memorial Hermann
Brief Title: Single Center Post Approval Proximal Humerus Fixation With the Conventus Cage PH™ Device
Status: Terminated | Type: Observational
Why Stopped: Study stopped due to business decision to not continue to gather clinical evidence on product
Sponsor: Conventus Orthopaedics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 7821
Record Dates: First submitted 2018-09-27; First posted 2018-10-18 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2019-09

CONDITIONS: Proximal Humeral Fracture
Keywords: Proximal humerus fracture fixation; Trauma; Proximal Humerus; Fixation
MeSH Terms: conditions — Shoulder Fractures; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Conventus Cage PH device — The Conventus CAGE™ PH (PH Cage) is a permanent implant comprised of an expandable scaffold, made from nitinol and titanium, which is deployed into the medullary canal and provides a structure to which fractured bone fragments are attached using fragment screws.

SUMMARY:
The Conventus CAGE™ PH (PH Cage) System Post-Approval Observational Data Collection Study (Study) is a single center, prospective, post-approval clinical study designed to collect device and procedure experience in everyday clinical practice.

DETAILED DESCRIPTION:
The study is a prospective, non-randomized, post-market approval data collection study that is designed to collect device/procedure and outcome data on patients who have experienced proximal humerus bone fractures and received a PH Cage.

Specifically, the study will provide:

1. Patient outcome and performance data for the implant and implant procedure that that may be used to support scientific publications.
2. Assurance of continued product safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be of at least legal age of consent according to applicable State Law.
* Patient is able to understand and provide written consent

Exclusion Criteria:

* The PH Cage should not be implanted in patients with suspected or known allergies to titanium or nickel.
* Pregnant female patients.
* Patients with current or history of mental illness and/or senility.
* Patients with current or history of alcoholism and/or chemical substance abuse.
* Patient has a medical condition(s) that preclude cooperation with the rehabilitation regimen.
* Patient has active infection at the operative site or other active systemic infection.
* Patient has a pathologic proximal humerus fracture.
* Patients proximal humerus fracture extends into the diaphysis.
* Patient has associated glenohumeral dislocation.
* Patient has known pre-existing rotator cuff disease.
* Patient has ipsilateral injury or concomitant surgery that will have a material impact on the study, such that the injury/surgery affects the patients' health status or the function of the injured extremity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled from the community in which the study is being conducted.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Primary Performance Patient Assessment | Change from Baseline in Constant Murley Score at the 2 year post op
  Constant Murley Score (CMS) The Constant Murley Score is a combination of visual analog scales assessing pain, activities of daily living and assessments of range of motion and strength using a long-armed goniometer and isometer. The higher the score the better for the following sections of the CMS: A. Pain (0-15 points) (e.g.15=no pain, 2=high pain), B. Everyday activities-question 1 (0-2 points) (e.g. 2=best, 0=worst), questions 2 and 3(0-4 points) (the higher the score the better), question 4 (0-10 points) C. Movement- questions 1 and 2 (0-20 points) (e.g. the greater the range of motion performed, the more points assigned), questions 3 and 4 (0-10 points) (e.g. points assigned based on movements performed) D. Strength (0-25 points) Score is calculated from the highest score of three attempts, with each score corresponding to the force in pounds (max 25 points) The overall score is then calculated by combining all sections (A+B+C+D= 0-100 points)

CONTACTS AND LOCATIONS:
Overall Officials: James M Gregory, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Carrie M Hill, Study Director — Conventus Orthopaedics, Inc.
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected will be used to support publications; all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: The data will become available once the study concludes (>2 years from date of first enrollment, until last patient followed) Data will be publicly available via any publications developed from this study. Length of availability will be determined by the publishing party.
Access Criteria: Data will be publicly available via any publications developed from this study.